CLINICAL TRIAL: NCT03600324
Title: Randomized Controlled Trial for Vestibular Treatment in Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PRO18070243; PT170144 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vestibular Disorder; Mild Traumatic Brain Injury
Keywords: mild traumatic brain injury; vestibular impairment; vestibular rehabilitation
MeSH Terms: conditions — Vestibular Diseases; Brain Concussion

STUDY DESIGN:
Intervention Model Description: A prospective, single-blind, four-group multi-center randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Intensity/Low Frequency (Experimental): Participants will be assigned T-REV with low intensity (30% of perceived effort) and low frequency (exercises performed 1x/day)
  Interventions: Behavioral: T-REV
- Low Intensity/ High Frequency (Experimental): Participants will be assigned T-REV with low intensity (30% of perceived effort) and high frequency (exercises performed 2x/day)
  Interventions: Behavioral: T-REV
- High Intensity/Low Frequency (Experimental): Participants will be assigned T-REV with high intensity (70% of perceived effort) and low frequency (exercises performed 1x/day)
  Interventions: Behavioral: T-REV
- High Intensity/High Frequency (Experimental): Participants will be assigned T-REV with high intensity (70% of perceived effort) and high frequency (exercises performed 2x/day)
  Interventions: Behavioral: T-REV

INTERVENTIONS:
Behavioral: T-REV — For any intervention that involves physical exercise, four parameters must be specified to complete the prescription; Type (mode), Intensity, Frequency, and Time. o The standard of care vestibular rehabilitation exercise program consists of three types of treatments that target the specific impairments and limitations discovered during the examination. The three types are: 1) gaze stabilization for vestibulo-ocular reflex dysfunction, 2) visual-vestibular habituation exercise for visual motion sensitivity, and 3) balance exercises for standing balance or gat dysfunction.

SUMMARY:
A prospective, single-blind, four-group multi-center randomized controlled trial (RCT) of targeted rehabilitation exercises for vestibular symptoms and impairments (T-REV) in civilians with mild traumatic brain injury (mTBI) will be conducted at the University of Pittsburgh Medical Center Sports Medicine Concussion Program (UPitt). The four treatment groups will consist of the factorial combinations of low (30%) and high (70%) intensity of exercise crossed with low (12-18 min, 1x/day) and high (12-18 min, 2x/day) frequency. A total of 125 participants aged 18-50 years will be enrolled across years 1-4, with approximately 100 participants completing the whole study. After potential participants with mTBI are screened for the vestibular clinical profile, using domain-specific tests and measures, and enrolled into the study, participants will complete primary and secondary outcome measures and receive a home exercise program that a) targets participants individual deficits, and b) is of the appropriate intensity and frequency for the participant's randomly assigned treatment group. Participants will return for in-clinic visits once per week to receive treatment and progress assigned exercises.

DETAILED DESCRIPTION:
During the past 17 years, US military personnel experienced 305,000 mTBI (DVBIC, 2017), with an estimated 65% (187,000) involving some type of vestibular impairment (gaze, postural/dynamic instability) and symptoms (dizziness, vertigo, motion intolerance) (Mucha et al., 2014). These vestibular impairments and symptoms, which have been associated with poor outcomes following mTBI including longer recovery times (Lau et al., 2011), can be actively treated using targeted vestibular rehabilitation exercises (Alsalaheen et al., 2010). In fact, the investigators recently concluded an observational trial of military personnel and civilians with mTBI- Targeted Evaluation, Action and Monitoring of TBI (TEAM-TBI) project (W81XWH-14-2-0002) supporting the effectiveness of targeted vestibular rehabilitation exercises in military personnel and civilians with complex mTBI (Kontos et al., in press). Although these vestibular-focused rehabilitation exercises are commonly used by military medical personnel following complex mTBI, there are no well-designed studies that show how much these exercises should be performed to be effective in US military personnel. In short, the concussion rehabilitation field does not know how frequently or intensely the exercises should be performed in order for injured personnel to have the best recovery.

In the current proposal, the investigators leverage our interdisciplinary team of experts from physical therapy, neurology, neuropsychology, and sports medicine and over 17 years of clinical and research experience to conduct a RCT comparing different frequency and intensity of targeted vestibular therapeutic exercises in military personnel and civilians. In so doing, the proposed study may inform a more precise approach for treating vestibular symptoms and impairments following mTBI that minimizes morbidity and accelerates recovery. Deliverables from the current study include: 1) outcome data regarding the efficacy of different frequencies and intensities of targeted vestibular exercises in both military personnel and civilians, and 2) evidence-based clinical practice guidelines (CPG) for prescribing vestibular therapeutic exercises.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Normal/corrected vision
* Diagnosed with sport-related mTBI/concussion in the past 8 days-1 year with clear mechanism of injury
* Glasgow coma scale (GCS) of 13 or greater
* Reported signs of mTBI including: loss of consciousness, amnesia, disorientation, confusion, dizziness, imbalance, memory problems, vomiting
* mTBI-related vestibular symptoms (dizziness, vertigo, motion intolerance) and/or impairments (gaze stabilization, standing balance, functional gait) per a comprehensive assessment, clinical exam, and interview

Exclusion Criteria:

* History of vestibular disorder prior to current mTBI (benign paroxysmal positional vertigo, unilateral or bilateral vestibular hypofunction)
* Benign Paroxysmal Positional Vertigo (BPPV) resulting from vestibular hypofunction
* Dizziness symptoms that only result from exercise
* History of neurological disorder
* <1 month or >6 months following current mTBI
* Currently pregnant or become pregnant during study
* Currently involved in litigation associated with current or previous mTBI Note: history of motion sickness/sensitivity will NOT be excluded. We will adjust for any imbalance in groups on this factor by covariate analysis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | enrollment, 2-week, 4-week, 3-month study visits
  The DHI is a 25-item self-report measure that examines dizziness-related handicap. Each item is categorized into one of three domains: functional, emotional, or physical. The DHI was developed with the help of patients who complained of dizziness and uses a three-item response scale (Yes, Sometimes, No) scored as 4/2/0, respectively. Score range: 0-100. The DHI has good internal consistency for the total score (alpha = 0.89). the test-retest reliability is high (r=0.97) and is response to change in a vestibular population. The DHI has been demonstrated to be valid in individuals with mTBI. The outcome measure will be assessed at multiple timepoints to assess change over time.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | enrollment, 2-week, 4-week, 3-month study visits
  The PGIC will be completed by all participants. The PGIC was developed for self-reported assessment of change resulting from post-concussion care at military treatment facilities. The prompt is: "Since beginning treatment at this facility, how would you describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life rated to your post-concussion condition?" The patient responds on a scale 0 (no change or condition has worsened) to 7 (considerable improvement). Because not all participants will have had a mTBI that precipitated the referral for physical therapy, the prompt will be modified to delete "post-concussive' for these cases. The interest for this measure is in the change between timepoints.
Neurobehavioral Symptom Inventory (NSI) | enrollment, 2-week, 4-week, 3-month study visits
  The NSI is a 22-item symptoms scale in which participants rate the severity of symptoms on a 5-point scale (0=none, 1= mild, 2=moderate, 3=severe, 4=very severe) Scores range from 0 to 60. The NSI takes approximately 5-10 minutes to administer. We are interested in the change in NSI over time.
Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) | enrollment, 2-week, 4-week study visits
  The ImPACT will be used to assess neurocognitive performance in civilians. ImPACT is a computerized neurocognitive test that includes six modules: 1) verbal memory, 2) design memory, 3) X's and O's, 4) symbol matching, 5) color matching, and 6) three letter memory. These modules are used to form four composite cores: verbal and visual memories (%), visual motor processing speed (#), and reaction time (sec). The ImPACT takes 20-30 minutes to administer. The interest in ImPACT scores is in both each timepoint to assess cognitive performance against the normal for age and change between time points as an assessment of recovery.
Pittsburgh Sleep Quality Index (PSQI) | enrollment, 2-week, 4-week study visits
  The PSQI will be used to assess sleep quality and consists of an 18-item self-report of seven component scores: 1) subjective sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disturbances, 6) sleep medication usage, and 7) daytime dysfunction. Scale for PSQI is 0 = not during past month; 1 = less than once a week; 2 = once or twice a week; 3 = three or more times a week. From the 18-item scores, seven component scores are calculated. A component score of 5 or greater is indicative of poor sleep quality. Sub-scale and global PSQI scores are calculated and higher scores indicating poorer sleep quality. The scores will be analyzed both at each timepoint to compare against normative values and between time points as an assessment of recovery.
Identify (ID) Migraine | enrollment, 2-week, 4-week study visits
  The ID Migraine is a 3-item screening tool designed to assess presence (yes/no) of symptoms related to headache/migraine pain including nausea, sensitivity to light, and functional impact of headaches. Scale for ID Migraine is 0 = no, 1 = yes. Scores range from 0-3 with clinical cut-off at 2 or greater indicating presences of migraine. The ID Migraine is both a valid and reliable screening tool for migraine with good combined sensitive and specificity. For the current study, we will adapt the ID Migraine tool by replacing the "during the last three months" time frame stem, with "following your injury". The ID Migraine requires 2 minutes to complete and score. he scores will be analyzed both at each timepoint to assess performance against clinical cutoffs and between time points as an assessment of recovery.
Neck Pain Numerical Rating Scale (Neck Pain NRS) | enrollment, 2-wk, 4-wk study visits
  The Defense and Veterans Pain Rating Scale (DVPRS) will be used specifically for neck pain. We will adapt the Defense and Veterans Pain Rating Scale (DVPRS) which was created to standardize pain reporting and measurement across the military. Changes to the verbal anchors include: 0 = "no pain", 1 = "hardly notice pain", 2 = "Notice pain, does not interfere with activities", 9 = "can't bear the pain, unable to do anything", 10 = "As bad as it could be, nothing else matters". Participants will be asked for their current neck pain during the past week. The Neck Pain NRS takes 1 minute to administer. The score will be analyzed both at each timepoint to assess current pain and compared over time to assess pain recovery.
Dizziness Numerical Rating Scale (Dizziness NRS) | enrollment, 2-wk, 4-wk study visits
  The Defense and Veterans Pain Rating Scale (DVPRS) will be used specifically for dizziness. We will adapt the Defense and Veterans Pain Rating Scale (DVPRS) which was created to standardize pain reporting and measurement across the military. Changes to the verbal anchors include: 0 = "no dizziness", 1 = "hardly notice dizziness", 2 = "Notice dizziness, does not interfere with activities", 9 = "can't bear the dizziness, unable to do anything", 10 = "As bad as it could be, nothing else matters". Participants will be asked for their current dizziness during the past week. The Dizziness NRS takes 1 minute to administer. The score will be analyzed both at each timepoint to assess current dizziness and compared over time to assess dizziness recovery.
Behavioral Symptom Inventory-18 (BSI-18) | enrollment, 2-week, 4-week study visits
  The BSI-18 is an 18-item symptom inventory that assesses the level of psychological distress during the past 7 days on 18 items. Symptoms are rated on a 5-point Likert scale ranging from 0 (not at all); 1 (a little bit); 2 (moderately); 3 (quite a bit); 4 (extremely). The BSI-18 yields total global severity index ranging from 0-72 as well as somatic, depression, and anxiety sub-scale scores. Any sub-scale T-score >63 is reflective of clinical impairment on that sub-scale. The BSI-18 requires 5 minutes to complete and score. Scores will be analyzed at each timepoint to assess current behavioral symptoms and impairments and compared over time to assess changes in symptoms.
Return to Activity (RTA) | 4-week, 3-month study visits
  Return to Activity will be medical clearance to resume full activities based on symptom and impairment free at rest, and symptom free following standardized exertion protocols per recent consensus. RTA will be assessed at 4 weeks and 3 months post-intervention.
International Physical Activity Questionnaire (IPAQ) | enrollment, 2-week, 4-week study visits
  The International Physical Activity Questionnaire (IPAQ) will assess potential treatment group difference in activity level. The IPAQ is a validated tool to assess recall of average activity level and intensity over the preceding 7 days. The IPAQ will be completed via text/online survey at 7 and 21 days and in person at 14 and 28 days during the clinic visits. The IPAQ was chosen because it is brief and can be either self-administered or administered via structured interview. Activity levels can be expressed as categorical variables (low, medium, high activity levels) or a continuous variable (MET-min/week). The IPAQ takes approximately 5 minutes to complete. Data will be analyzed at each timepoint and over time to assess changes in physical activity.
Visual Vertigo Analog Scale (VVAS) | 2-week, 4-week study visits
  The VVAS assesses how much dizziness 0 (none) to 10 (severe), on a visual analog scale, an individual reports for 9 different activities, such as walking through a supermarket aisle, being in a room with fluorescent lights, doing down and escalator, walking over a patterned floor, etc. A positive result occurs when an individual rates at least two of the nine items of the VVAS above zero (VVAS positive). The VVAS takes 5 minutes to administer. We will assess VVAS data at each timepoint and over time.
Vestibular Ocular Motor Screening (VOMS) | 2-wk, 4-wk study visits
  The VOMS assesses impairment via patient-reported symptom provocation following each of the following components: 1) smooth pursuits; 2) horizontal and vertical saccades; 3) convergence; 4) horizontal and vertical ocular reflex (VOR); and 5) visual motion sensitivity (VMS). Patients rate changes in headache, dizziness, nausea, and fogginess compared to their immediate pre-assessment state on a scale of 0 (none) to 10 (severe) to determine if any domain provokes symptoms. Scores on any VOMS item of 2 or greater reflects a positive screening cut-off for vestibular or oculomotor impairment. Convergence is also assessed in the VOMS using both symptom report and objective measurement of the near point of convergence (NPC, averaged across 3 trials). NPC values >5 cm reflect a positive clinical metronome, and a 1-page scoring form. The VOMS requires 5 minutes to administer and score. We will analyze VOMS at each timepoint and over time.
Modified Balance Error Scoring System (mBESS) | 2-week, 4-week study visits
  The mBESS measures postural stability and consists of three stances including feet side by side, a tandem stance, and a single-leg stance on the non-dominant leg. The three stances are performed for 20 seconds each on a firm surface. All stances are completed with eyes closed and with hands on the iliac crests. Errors include lifting hands off the iliac crests, opening the eyes, stepping, stumbling, falling, moving the hips more than 30 degrees of flexion or abduction, lifting the forefoot or heel, or remaining out of the testing position for more than 5 seconds. Each error equals 1 point, with higher scores indicating worse performance. For the current study, we will use the modified BESS (mBESS) on the firm surface only. Clinical cut-offs for BESS suggest a total error of 9 or greater indicate clinical impairment in balance. The mBESS takes approximately 5-6 minutes to administer. mBESS scores will be analyzed at each timepoint and over time.
Functional Gait Assessment (FGA) | enrollment, 2-week, 4-week study visits
  FGA is 10 items that assess ability of participants to walk with head turns, changes of speed, and around obstacles. Each item is scored on a 4-point ordinal scale ranging from 0 (severe) to 3 (normal). Higher scores indicate normal gait.
High Level Mobility Assessment Tool (HiMAT) | enrollment, 2-week, 4-week study visits
  Assess balance, participants will complete only 1 subtest of the HiMAT, fast walking.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Kontos, PhD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Warrior Recovery Center, Colorado Springs, Colorado
  - Naval Medical Center Camp Lejeune - Intrepid Spirit Concussion Recovery Center, Marine Corps Base Camp Lejeune, North Carolina
  - UPMC/Univ of Pgh Sports Medicine Concussion Research Program, Pittsburgh, Pennsylvania
  - Carl R. Darnall Army Medical Center - Intrepid Spirit Center, Fort Hood, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers. For all study presentations and reports, aggregate data will be published.